CLINICAL TRIAL: NCT00925587
Title: A Multicenter, Randomised, Double-Blind Study Comparing De Novo Once Monthly and Once Every 2 Week Darbepoetin Alfa Dosing for the Correction of Anemia in Subjects With Chronic Kidney Disease Not Receiving Dialysis
Brief Title: Evaluation of Monthly Darbepoetin Alfa Dosing for Correction of Anemia in Non-dialysis Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20060163; 2006-003173-27 (EudraCT Number)
Record Dates: First submitted 2009-05-28; First posted 2009-06-22 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: CKD; Anemia; correction; darbepoetin alfa
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Q2W (Active Comparator): Q2W administration of darbepoetin alfa.
  Interventions: Drug: darbepoetin alfa
- QM (Active Comparator): QM administration of darbepoetin alfa
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa — Drug administered either Q2W or QM using a prefilled syringe. Allowable doses of: 10, 20, 30, 40, 50, 60, 80, 100, 130, 150, 200, 300, 400 or 600 mcg.
  Other Names: Placebo

SUMMARY:
The purpose of this study is to determine whether once monthly (QM) dosing of darbepoetin alfa is non-inferior to that of once every 2 week (Q2W) dosing of darbepoetin alfa for the correction of anemia in patients with Chronic Kidney Disease who are not receiving dialysis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosis of chronic kidney disease with eGFR of 15-59 mL/min/1.73 m2 (MDRD equation)
* Two consecutive screening Hb values taken at least 7 days apart must each be <10.0 g/dL
* TSAT ≥ 15%

Exclusion Criteria:

* Upper or lower GI bleeding within 6 months before enrolment
* ESA use within 12 weeks before enrolment
* Uncontrolled hypertension
* Systemic haematologic disorders
* Prior history within 12 weeks before enrollment of events including: Acute myocardial ischemia, unstable angina, myocardial infarction, hospitalization for congestive heart failure, stroke or transient ischaemic attack, limb ischaemia, deep vein thrombosis, thromboembolism.
* Grand mal seizure within 6 months prior to enrolment
* Evidence of, or received chemotherapy or radiation therapy for, a malignancy within 5 years prior to enrolment.
* Red blood cell transfusion within 12 weeks prior to enrolment
* Androgen therapy within 8 weeks prior to enrolment
* Pregnancy or breast feeding, or inadequate contraception
* Currently receiving immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2009-06; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (138):
- Australia (9):
  - Research Site, Gosford, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, New Lambton, New South Wales
  - Research Site, Randwick, New South Wales
  - Research Site, Cairns, Queensland
  - Research Site, Box Hill, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Reservoir, Victoria
- Belgium (6):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, LiÃ¨ge
  - Research Site, Roeselare
- Bulgaria (3):
  - Research Site, Pleven
  - Research Site, Sofia
  - Research Site, Varna
- Czechia (12):
  - Research Site, Brno
  - Research Site, Chrudim
  - Research Site, Jilemnice
  - Research Site, Kladno
  - Research Site, Liberec
  - Research Site, Nový Jičín
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Praha 4 - Nusle
  - Research Site, Slavkov u Brna
  - Research Site, Sternberk
  - Research Site, Ústí nad Orlicí
- Denmark (3):
  - Research Site, Ã…rhus
  - Research Site, Roskilde
  - Research Site, Viborg
- Research Site, Tallinn, Estonia
- France (10):
  - Research Site, Annonay
  - Research Site, Creil
  - Research Site, Grenoble
  - Research Site, Metz
  - Research Site, Montivilliers
  - Research Site, Nice
  - Research Site, Poissy
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Saint-Priest-en-Jarez
- Germany (5):
  - Research Site, Bernkastel-Kues
  - Research Site, Coesfeld
  - Research Site, DÃ¼sseldorf
  - Research Site, Hamburg
  - Research Site, Leverkusen
- Greece (4):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Larissa
  - Research Site, Thessaloniki
- Hungary (10):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Esztergom
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Pécs
  - Research Site, Szekszárd
  - Research Site, Szombathely
  - Research Site, Zalaegerszeg
- Israel (3):
  - Research Site, Ashkelon
  - Research Site, Hadera
  - Research Site, Jerusalem
- Italy (9):
  - Research Site, Albano Laziale RM
  - Research Site, Ancona
  - Research Site, Cagliari
  - Research Site, Florence
  - Research Site, Lecco
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Torino
- Latvia (4):
  - Research Site, Daugavpils
  - Research Site, Riga
  - Research Site, Valmiera
  - Research Site, Ventspils
- Mexico (5):
  - Research Site, Saltillo, Coahuila
  - Research Site, Guadalajara, Jalisco
  - Research Site, Cuernavaca, Morelos
  - Research Site, Querétaro, QuerÃ©taro
  - Research Site, San Luis Potosí City, San Luis PotosÃ-
- Poland (10):
  - Research Site, Choszczno
  - Research Site, Golub-Dobrzyń
  - Research Site, Koszalin
  - Research Site, Kościerzyna
  - Research Site, Legnica
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Zamość
- Portugal (5):
  - Research Site, Evora
  - Research Site, Faro
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, SetÃºbal
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Timișoara
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yekaterinburg
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Krgujevac
  - Research Site, Zemun
- Slovakia (6):
  - Research Site, Bratislava
  - Research Site, Galanta
  - Research Site, Námestovo
  - Research Site, Šaľa
  - Research Site, Trstená
  - Research Site, Zvolen
- Slovenia (4):
  - Research Site, Jesenice
  - Research Site, Novo Mesto
  - Research Site, Slovenj Gradec
  - Research Site, Šempeter pri Gorici
- Spain (6):
  - Research Site, JaÃ©n, AndalucÃ-a
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, L'Hospitalet de Llobregat, CataluÃ±a
  - Research Site, Madrid, Madrid
  - Research Site, Majadahonda, Madrid
  - Research Site, Galdakao, PaÃ-s Vasco
- United Kingdom (14):
  - Research Site, Birmingham
  - Research Site, Brighton
  - Research Site, Cambridge
  - Research Site, Coventry
  - Research Site, Glasgow
  - Research Site, Hull
  - Research Site, Leicester
  - Research Site, Newcastle upon Tyne
  - Research Site, Salford
  - Research Site, Shrewsbury
  - Research Site, Stevenage
  - Research Site, Stoke-on-Trent
  - Research Site, Swansea
  - Research Site, Wolverhampton

REFERENCES:
- [Derived] Roger SD, Kolmakova E, Fung M, Malecki R, Vinhas J, Dellanna F, Thomas M, Manamley N, Ferenczi S. Darbepoetin alfa once monthly corrects anaemia in patients with chronic kidney disease not on dialysis. Nephrology (Carlton). 2014 May;19(5):266-74. doi: 10.1111/nep.12214. PMID 24506498
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Darbepoetin Alfa Q2W: Darbepoetin alfa Intravenous Once Every 2 Weeks
- Darbepoetin Alfa QM: Darbepoetin alfa Intravenous Once Monthly
Period: Overall Study
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Started | 178 | 180
Completed | 142 | 155
Not Completed | 36 | 25
Not completed — Protocol Specified Criteria | 6 | 6
Not completed — Physician Decision | 4 | 1
Not completed — Protocol Violation | 6 | 4
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Death | 5 | 5
Not completed — Adverse Event | 6 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Includes all subjects who received at least one dose of darbepoetin alfa on study. 3 subjects randomized to the Q2W arm failed to administer darbepoetin alfa
Groups:
- Total: Total of all reporting groups
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM | Total
Number analyzed (Participants) | 175 | 180 | 355
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (14.1) | 66.3 (15.2) | 67.3 (14.7)
Age, Customized [Number; unit: Participants]
  <65 years | 60 | 67 | 127
  >=65-<75 years | 42 | 54 | 96
  >=75 years | 73 | 59 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 104 | 211
  Male | 68 | 76 | 144
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 0 | 1 | 1
  White or Caucasian | 166 | 163 | 329
  Other | 9 | 16 | 25
Baseline Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 9.13 (0.61) | 9.11 (0.70) | 9.12 (0.65)

OUTCOME MEASURES:

1. Primary Outcome: Hb Change Between Baseline and the Evaluation Period (Average of Weeks 29-33)
Description: The Adjusted Analysis is the primary analysis and includes treatment group and baseline Hb value as covariates. Non-inferiority is concluded if the lower limit of the 95% confidence interval for the mean difference is above -0.5g/dL.
Time Frame: Baseline Week 33
Population: Primary Analysis Set: All subjects receiving at least one dose of darbepoetin alfa in the treatment group to which they were randomized and with at least one evaluable (not within 90 days after an RBC transfusion) Hb measurement during the evaluation period (Weeks 29-33)
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 154
g/dL | 2.157 [1.984 to 2.330] | 1.969 [1.803 to 2.135]
Statistical Analysis 1: Comparison: Darbepoetin Alfa Q2W vs Darbepoetin Alfa QM; Power = 90% at sample size calculation; Test type: Non-Inferiority or Equivalence — Non-inferiority margin -0.5 g/dL; Mean Difference (Final Values) = -0.188, 95% CI 2-sided [-0.427 to 0.052], Standard Error of Mean 0.122 — Darbepoetin alfa QM - Darbepoetin alfa Q2W

2. Secondary Outcome: Achievement of Both a Hb >= 10.0 g/dL and a >= 1.0 g/dL Increase From Baseline at Any Time Point Following de Novo Darbepoetin Alfa Administration.
Time Frame: Baseline to Week 33
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 154
Percentage of Participants | 97.9 [95.5 to 100.0] | 98.1 [95.9 to 100.0]

3. Secondary Outcome: Hb at Baseline
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 154
g/dL | 9.17 (0.05) | 9.12 (0.06)

4. Secondary Outcome: Hb at Week 3
Time Frame: Week 3
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 153
g/dL | 9.89 (0.08) | 10.13 (0.10)

5. Secondary Outcome: Hb at Week 5
Time Frame: Week 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 152
g/dL | 10.58 (0.08) | 10.28 (0.09)

6. Secondary Outcome: Hb at Week 7
Time Frame: Week 7
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 140 | 152
g/dL | 10.90 (0.09) | 10.75 (0.10)

7. Secondary Outcome: Hb at Week 9
Time Frame: Week 9
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 140 | 153
g/dL | 11.24 (0.10) | 10.79 (0.10)

8. Secondary Outcome: Hb at Week 11
Time Frame: Week 11
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 151
g/dL | 11.35 (0.10) | 11.17 (0.10)

9. Secondary Outcome: Hb at Week 13
Time Frame: Week 13
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 140 | 149
g/dL | 11.56 (0.10) | 11.05 (0.10)

10. Secondary Outcome: Hb at Week 15
Time Frame: Week 15
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 150
g/dL | 11.42 (0.11) | 11.25 (0.09)

11. Secondary Outcome: Hb at Week 17
Time Frame: Week 17
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 138 | 150
g/dL | 11.66 (0.10) | 11.12 (0.09)

12. Secondary Outcome: Hb at Week 19
Time Frame: Week 19
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 148
g/dL | 11.50 (0.12) | 11.20 (0.09)

13. Secondary Outcome: Hb at Week 21
Time Frame: Week 21
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 137 | 146
g/dL | 11.53 (0.10) | 11.09 (0.08)

14. Secondary Outcome: Hb at Week 23
Time Frame: Week 23
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 138 | 148
g/dL | 11.36 (0.09) | 11.08 (0.09)

15. Secondary Outcome: Hb at Week 25
Time Frame: Week 25
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 151
g/dL | 11.34 (0.10) | 10.85 (0.09)

16. Secondary Outcome: Hb at Week 27
Time Frame: Week 27
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 138 | 150
g/dL | 11.22 (0.09) | 11.07 (0.09)

17. Secondary Outcome: Hb at Week 29
Time Frame: Week 29
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 137 | 151
g/dL | 11.35 (0.10) | 10.90 (0.09)

18. Secondary Outcome: Hb at Week 31
Time Frame: Week 31
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 140 | 152
g/dL | 11.31 (0.09) | 11.28 (0.09)

19. Secondary Outcome: Hb at Week 33
Time Frame: Week 33
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 136 | 149
g/dL | 11.38 (0.10) | 11.15 (0.10)

20. Secondary Outcome: Darbepoetin Alfa Dose at Week 1
Description: Although the endpoint is related to dose, the sample is from the Primary Analysis Set which requires a Hb value in the evaluation period
Time Frame: Week 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 154
µg/wk | 27.65 (0.10) [26.59 to 28.76] | 27.06 (0.10) [26.09 to 28.06]

21. Secondary Outcome: Darbepoetin Alfa Dose at Week 3
Description: as for outcome 20
Time Frame: Week 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 154
µg/wk | 25.80 (0.10) [24.64 to 27.00] | 27.06 (0.10) [26.09 to 28.06]

22. Secondary Outcome: Darbepoetin Alfa Dose at Week 5
Description: as for outcome 20
Time Frame: Week 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 153
µg/wk | 24.40 (0.10) [22.70 to 26.23] | 24.52 (0.10) [22.70 to 26.50]

23. Secondary Outcome: Darbepoetin Alfa Dose at Week 7
Description: as for outcome 20
Time Frame: Week 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 153
µg/wk | 23.42 (0.10) [21.42 to 25.61] | 24.52 (0.10) [22.70 to 26.50]

24. Secondary Outcome: Darbepoetin Alfa Dose at Week 9
Description: as for outcome 20
Time Frame: Week 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 154
µg/wk | 20.01 (0.10) [17.36 to 23.07] | 20.59 (0.10) [17.89 to 23.70]

25. Secondary Outcome: Darbepoetin Alfa Dose at Week 11
Description: as for outcome 20
Time Frame: Week 11
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 154
µg/wk | 18.99 (0.10) [16.22 to 22.24] | 20.50 (0.10) [17.83 to 23.58]

26. Secondary Outcome: Darbepoetin Alfa Dose at Week 13
Description: as for outcome 20
Time Frame: Week 13
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 151
µg/wk | 14.67 (0.10) [11.97 to 17.98] | 19.52 (0.10) [16.79 to 22.69]

27. Secondary Outcome: Darbepoetin Alfa Dose at Week 15
Description: as for outcome 20
Time Frame: Week 15
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 153
µg/wk | 14.19 (0.10) [11.52 to 17.47] | 19.15 (0.10) [16.42 to 22.33]

28. Secondary Outcome: Darbepoetin Alfa Dose at Week 17
Description: as for outcome 20
Time Frame: Week 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 140 | 153
µg/wk | 12.71 (0.10) [10.15 to 15.92] | 19.94 (0.10) [17.28 to 23.02]

29. Secondary Outcome: Darbepoetin Alfa Dose at Week 19
Description: as for outcome 20
Time Frame: Week 19
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 153
µg/wk | 14.52 (0.10) [11.97 to 17.61] | 19.94 (0.10) [17.28 to 23.01]

30. Secondary Outcome: Darbepoetin Alfa Dose at Week 21
Description: as for outcome 20
Time Frame: Week 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 140 | 150
µg/wk | 15.42 (0.10) [12.96 to 18.36] | 21.59 (0.10) [19.20 to 24.29]

31. Secondary Outcome: Darbepoetin Alfa Dose at Week 23
Description: as for outcome 20
Time Frame: Week 23
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 154
µg/wk | 14.73 (0.10) [12.35 to 17.57] | 19.98 (0.10) [17.39 to 22.94]

32. Secondary Outcome: Darbepoetin Alfa Dose at Week 25
Description: as for outcome 20
Time Frame: Week 25
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 153
µg/wk | 14.55 (0.10) [12.16 to 17.41] | 20.70 (0.10) [18.10 to 23.68]

33. Secondary Outcome: Darbepoetin Alfa Dose at Week 27
Description: as for outcome 20
Time Frame: Week 27
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 154
µg/wk | 16.07 (0.10) [13.69 to 18.85] | 20.79 (0.10) [18.18 to 23.77]

34. Secondary Outcome: Darbepoetin Alfa Dose at Week 29
Description: as for outcome 20
Time Frame: Week 29
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 137 | 151
µg/wk | 15.06 (0.10) [12.75 to 17.78] | 20.57 (0.10) [17.74 to 23.85]

35. Secondary Outcome: Darbepoetin Alfa Dose at Week 31
Description: as for outcome 20
Time Frame: Week 31
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 153
µg/wk | 14.48 (0.10) [12.20 to 17.19] | 19.39 (0.10) [16.51 to 22.77]

36. Secondary Outcome: Darbepoetin Alfa Dose During the Evaluation Period (Average of Weeks 29-33)
Description: as for outcome 20
Time Frame: Weeks 29-33
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 140 | 153
µg/wk | 15.21 (0.10) [12.99 to 17.81] | 19.68 (0.10) [16.84 to 23.01]

37. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 3
Description: as for outcome 20
Time Frame: Week 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 154
ratio | 0.931 (0.10) [0.914 to 0.947] | 1.000 (0.10) [1.000 to 1.000]

38. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 5
Description: as for outcome 20
Time Frame: Week 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 153
ratio | 0.882 (0.10) [0.832 to 0.936] | 0.907 (0.10) [0.845 to 0.974]

39. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 7
Description: as for outcome 20
Time Frame: Week 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 153
ratio | 0.845 (0.10) [0.782 to 0.914] | 0.907 (0.10) [0.845 to 0.974]

40. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 9
Description: as for outcome 20
Time Frame: Week 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 154
ratio | 0.724 (0.10) [0.631 to 0.832] | 0.761 (0.10) [0.662 to 0.875]

41. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 11
Description: as for outcome 20
Time Frame: Week 11
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 154
ratio | 0.684 (0.10) [0.588 to 0.797] | 0.758 (0.10) [0.659 to 0.871]

42. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 13
Description: as for outcome 20
Time Frame: Week 13
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 151
ratio | 0.531 (0.10) [0.435 to 0.647] | 0.719 (0.10) [0.620 to 0.835]

43. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 15
Description: as for outcome 20
Time Frame: Week 15
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 153
ratio | 0.512 (0.10) [0.417 to 0.628] | 0.707 (0.10) [0.608 to 0.823]

44. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 17
Description: as for outcome 20
Time Frame: Week 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 140 | 153
ratio | 0.459 (0.10) [0.368 to 0.572] | 0.737 (0.10) [0.641 to 0.847]

45. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 19
Description: as for outcome 20
Time Frame: Week 19
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 153
ratio | 0.525 (0.10) [0.435 to 0.633] | 0.737 (0.10) [0.641 to 0.846]

46. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 21
Description: as for outcome 20
Time Frame: Week 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 140 | 150
ratio | 0.556 (0.10) [0.471 to 0.656] | 0.797 (0.10) [0.713 to 0.891]

47. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 23
Description: as for outcome 20
Time Frame: Week 23
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 141 | 154
ratio | 0.533 (0.10) [0.450 to 0.632] | 0.738 (0.10) [0.646 to 0.844]

48. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 25
Description: as for outcome 20
Time Frame: Week 25
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 153
ratio | 0.526 (0.10) [0.443 to 0.625] | 0.764 (0.10) [0.671 to 0.869]

49. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 27
Description: as for outcome 20
Time Frame: Week 27
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 154
ratio | 0.581 (0.10) [0.499 to 0.677] | 0.768 (0.10) [0.675 to 0.875]

50. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 29
Description: as for outcome 20
Time Frame: Week 29
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 137 | 151
ratio | 0.544 (0.10) [0.462 to 0.640] | 0.762 (0.10) [0.661 to 0.880]

51. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at Week 31
Description: as for outcome 20
Time Frame: Week 31
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 153
ratio | 0.525 (0.10) [0.443 to 0.622] | 0.717 (0.10) [0.613 to 0.839]

52. Secondary Outcome: Dose of Darbepoetin Alfa at the First Achievement of a Hb ≥10.0 g/dL and a ≥1.0 g/dL Increase From Baseline (Weeks 1-33)
Description: as for outcome 20
Time Frame: Weeks 1-33
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/wk
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 139 | 151
µg/wk | 25.95 (0.10) [24.43 to 27.56] | 29.65 (0.10) [27.89 to 31.52]

53. Secondary Outcome: Time to First Achievement of a Hb ≥10.0 g/dL and a ≥1.0 g/dL Increase From Baseline (Weeks 1-33)
Time Frame: Weeks 1-33
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 142 | 154
Weeks | 5.0 [3.0 to 7.0] | 5.0 [3.0 to 9.0]

54. Secondary Outcome: Ratio of Darbepoetin Alfa Dose to Baseline at the Evalaution Period (Average of Weeks 29-33)
Description: as for outcome 20
Time Frame: Evaluation Period
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Number analyzed (Participants) | 140 | 153
ratio | 0.550 (0.10) [0.471 to 0.643] | 0.728 (0.10) [0.625 to 0.849]

ADVERSE EVENTS:
Time Frame: 33 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  Summary of Adverse Events includes only those subjects who received at least one dose of investigational product.
Arm/Group | Darbepoetin Alfa Q2W | Darbepoetin Alfa QM
Serious Adverse Events (participants affected / at risk) | 52/175 | 54/180
Other Adverse Events (participants affected / at risk) | 68/175 | 63/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa Q2W (N=175) | Darbepoetin Alfa QM (N=180)
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 6 | 3
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 3
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Generalised oedema (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 1
Spinal pain (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 1
Nephropathy (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 4 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 4
Renal failure chronic (Renal and urinary disorders) | 7 | 4
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 1 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa Q2W (N=175) | Darbepoetin Alfa QM (N=180)
Diarrhoea (Gastrointestinal disorders) | 10 | 7
Asthenia (General disorders) | 10 | 5
Oedema peripheral (General disorders) | 17 | 14
Urinary tract infection (Infections and infestations) | 8 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 12
Hypertension (Vascular disorders) | 36 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.